CLINICAL TRIAL: NCT01264562
Title: Cognition in Breast Cancer Patients: The Impact of Cancer-related Stress
Acronym: Cognicares
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Principal Investigator, Kerstin Hermelink, Study Principal Investigator, Ludwig-Maximilians - University of Munich
Other Study IDs: DKH 109132
Record Dates: First submitted 2010-12-20; First posted 2010-12-22 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Breast Cancer
Keywords: chemotherapy, adjuvant; adverse effects; breast neoplasms; cognition disorders; Stress Disorders, post-traumatic; cortisol
MeSH Terms: conditions — Breast Neoplasms; Cognition Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Chemotherapy group: Breast cancer patients treated with chemotherapy
- Non-chemotherapy group: Breast cancer patients not treated with chemotherapy
- Healthy controls: Women without a cancer diagnosis, matched for age and education

SUMMARY:
The study will investigate the impact of cancer-related stress and its consequences (acute and posttraumatic stress symptoms, altered cortisol secretion) on cognitive function in breast cancer patients. The hypothesis that stress associated with the cancer diagnosis and the cancer treatment is a major cause of cognitive dysfunction in breast cancer patients shall be evaluated.

DETAILED DESCRIPTION:
Primary hypothesis:

*The adverse effects of cancer and cancer therapy on cognitive function in breast cancer patients are entirely or partly mediated by stress and the ensuing dysfunction of the HPA-axis.

Secondary objectives:

* Determining the effect of cancer diagnosis, chemotherapy, disease-related stress, acute stress response, posttraumatic stress disorder, posttraumatic stress symptoms, anxiety, and depression on the HPA-axis in breast cancer patients
* Determining the effect of cognitive dysfunction assessed with neuropsychological tests, cancer diagnosis, chemotherapy, disease-related stress, acute stress response, posttraumatic stress disorder, posttraumatic stress symptoms, anxiety, and depression on subjective cognitive function in breast cancer patients
* Prevalence of acute stress response, posttraumatic stress disorder and posttraumatic stress symptoms, and extent of cancer-specific stress in breast cancer patients treated with or without chemotherapy

ELIGIBILITY:
Inclusion Criteria, both patient groups:

* primary breast cancer, stage 0-IIIc, therapy not yet started
* informed consent

Inclusion Criteria, healthy control group:

* breast diagnostics with benign result (no treatment necessary)
* informed consent

Exclusion Criteria:

* not fluent in German
* substance abuse
* history of psychosis
* history of neurologic disorder
* previous systemic cancer treatment
* Addison' disease
* Cushing's syndrome

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the Ludwig Maximilian University of Munich Breast Cancer Center; Klinikum Landshut Department of Obstetrics and Gynecology and Breast Cancer Services; Kreisklinik Ebersberg Department of Gynecology and Obstetrics; Klinikum Dritter Orden Department of Gynecology and Obstetrics; Rotkreuzklinikum Muenchen Department of Gynecology and Obstetrics, Helios Amper Hospital Dachau, Department of Gynecology and Obstetrics
Sampling Method: Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2011-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Course of cognitive function | 12 months
  Performance on a battery of cognitive tests

SECONDARY OUTCOMES:
Course of subjective cognitive function | 12 months
  Self-reported cognitive problems
Course of the HPA-axis function | 12 months
  Cortisol awakening response and diurnal profile
Course of the stress response | 12 months
  Acute stress response, posttraumatic stress disorder, and posttraumatic stress symptoms; cancer-specific stress

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin Hermelink, PhD, Principal Investigator — Ludwig Maximilian University, Department of Gynecology and Obstetrics
Locations (6):
- Germany (6):
  - Frauenklinik des Helios Amper Klinikums Dachau, Dachau, Bavaria
  - Kreisklinik Ebersberg, Ebersberg, Bavaria
  - Klinikum Landshut, Department of Obstetrics and Gynecology and Breast Cancer Services, Landshut, Bavaria
  - Rotkreuzklinikum Muenchen, Munich, Bavaria
  - Klinikum Dritter Orden, Munich, Bavaria
  - Ludwig Maximilian University, Department of Gynecology and Obstetrics, Munich, Bavaria

REFERENCES:
- [Background] Hermelink K, Buhner M, Harbeck N. Response. J Natl Cancer Inst. 2016 Apr 13;108(8):djw049. doi: 10.1093/jnci/djw049. Print 2016 Aug. No abstract available. PMID 27075856
- [Result] Hermelink K, Voigt V, Kaste J, Neufeld F, Wuerstlein R, Buhner M, Munzel K, Rjosk-Dendorfer D, Grandl S, Braun M, von Koch FE, Hartl K, Hasmuller S, Bauerfeind I, Debus G, Herschbach P, Harbeck N. Elucidating pretreatment cognitive impairment in breast cancer patients: the impact of cancer-related post-traumatic stress. J Natl Cancer Inst. 2015 Apr 16;107(7):djv099. doi: 10.1093/jnci/djv099. Print 2015 Jul. PMID 25882713
- [Result] Voigt V, Neufeld F, Kaste J, Buhner M, Sckopke P, Wuerstlein R, Hellerhoff K, Sztrokay-Gaul A, Braun M, von Koch FE, Silva-Zurcher E, Hasmuller S, Bauerfeind I, Debus G, Herschbach P, Mahner S, Harbeck N, Hermelink K. Clinically assessed posttraumatic stress in patients with breast cancer during the first year after diagnosis in the prospective, longitudinal, controlled COGNICARES study. Psychooncology. 2017 Jan;26(1):74-80. doi: 10.1002/pon.4102. Epub 2016 Feb 22. PMID 26898732
- See also: website of the Ludwig Maximilian University of Munich, Breast Cancer Center, Psycho-Oncology — http://www.klinikum.uni-muenchen.de/Brustzentrum/de/psychoonko/psy_grh/index.html